CLINICAL TRIAL: NCT03871764
Title: Relation of 3rd Trimester Uterine Artery Doppler Flow Velocimetry Indices, Factor V Leiden Mutation and Placental Pathology to the Severity of Preeclampsia
Brief Title: Prediction of Outcome in Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Nooh Riad Ali, professor, Cairo University
Other Study IDs: 019002
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Leiden Factor V Deficiency,Preeclampsia; Doppler Examination; Palental Pathology
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — blood samples and placental pathology
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood sample , doppler of uterine vessel and placenta — blood sample for factor V and doppler examination of uterine arteries , placenta pathology post partum

SUMMARY:
this summary studied the predictive values of factor V Leiden mutation , doppler indices , placental pathology to unfavorable fetal and maternal outcomes

DETAILED DESCRIPTION:
leiden mutation is activated protein C resistance with hypercoagulable states and increased thrombotic risk. 99 % are heterozygous and 1 % is homozygous , very rare cases are psoudohomozygous with factor V deficiency. relation to this mutation was studied in severe preeclamptic patients. doppler indices of uterine arteries , increased pulsetility index or unilateral or bilateral uterine artery notch and placental pathology were studied.

ELIGIBILITY:
Inclusion Criteria: severe preeclampsia in 3rd trimester -

Exclusion Criteria:Twin pregnancy. Fetal congenital anomalies. Diabetic patient, impaired renal function. Any medical disorders even that HTN. Any placental pathology,Autoimmune diseases. Women with uterine activity or clinical emergencies with maternal hemodynamic instability or an indication for immediate termination of pregnancy.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with preeclampsia in 3rd trimester. Singleton pregnancy. Accurate gestational age confirmed by last menstrual period or sonography before 20 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
percentage of patients develop abruption placenta, intrauterine growth retardation or delivered premature | within 12 wks from diagnosis of severe preeclampsia
  placental abruption, prematurity, IUGR
percentage of fetuses and neonates complicated with intrauterine fetal death or need admission to incubator | from diagnosis of severe preeclampsia till one week after delivery
  IUFD, admission to neonatal IUC

IPD SHARING:
Plan to Share IPD: No